CLINICAL TRIAL: NCT00020904
Title: A Phase II Study of Epothilone B Analog BMS-247550 in Patients With Taxane-Resistant Metastatic Breast Cancer
Brief Title: BMS-247550 in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-031; CDR0000068729 (Registry Identifier: PDQ (Physician Data Query)); BMS-CA163-009; CPMC-IRB-13916; NCI-G01-1967
Record Dates: First submitted 2001-07-11; First posted 2003-09-10 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating women who have stage IV or recurrent metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical activity of BMS-247550, in terms of tumor response rate, in women with taxane-resistant metastatic breast cancer.
* Determine the safety of this drug in these patients.
* Determine the duration of response, time to progression, and survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 3 hours on day 1. Treatment continues every 3 weeks for 4-18 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 4 additional courses beyond CR. Responding patients may receive additional courses at the investigator's discretion.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 14-50 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic breast carcinoma

  * Stage IV or recurrent disease with distant metastases
* Most recent prior chemotherapy was docetaxel-based or paclitaxel-based therapy for metastatic disease

  * Progressed during therapy or within 4 months of last dose OR
  * Progressed during therapy or within 6 months of last dose if given as adjuvant treatment only
* Received prior anthracycline therapy
* Bidimensionally measurable metastatic lesion

  * Bony lesions not considered measurable
* No known brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Sex:

* Female

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count greater than 125,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN (5 times ULN if hepatic metastases are present)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No unstable angina, myocardial infarction, or congestive heart failure within the past 6 months

Other:

* No grade 2 or greater neuropathy (motor or sensory)
* No uncontrolled infection or other medical illness that would preclude study
* No psychiatric disorder or other condition that would preclude study
* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No hypersensitivity to agents containing Cremophor EL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 24 hours since prior growth factor
* No concurrent trastuzumab (Herceptin)
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen for metastatic disease except an anthracycline-containing regimen as first-line therapy and a taxane as second-line therapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy (except hormone replacement therapy)

Radiotherapy:

* At least 3 weeks since prior radiotherapy, except palliative radiotherapy to less than 20% of the bone marrow, and recovered
* No prior radiotherapy to major bone marrow-containing areas (pelvis and lumbar spine)
* No prior radiotherapy to target lesion if only measurable lesion
* No concurrent therapeutic radiotherapy

Surgery:

* At least 1 week since prior minor surgery
* At least 3 weeks since prior major surgery
* Recovered from prior surgery

Other:

* Recovered from all prior treatment-related toxic effects (alopecia allowed)
* No other concurrent experimental anticancer medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A. Hudis, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York